CLINICAL TRIAL: NCT00985465
Title: Safety, Reactogenicity and Immunogenicity Study of GSK Biologicals' Pneumococcal Vaccine GSK1024850A, Given Either as a Booster Dose or as a 2-dose Catch-up Immunization in Healthy Malian Children
Brief Title: Immunization of Children Previously Primed With GSK Pneumococcal Vaccine GSK1024850A and of Unprimed Children in Mali
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 113166
Record Dates: First submitted 2009-09-24; First posted 2009-09-28 (Estimated); Results first posted 2018-12-14 (Actual); Last update posted 2018-12-14 (Actual); Status verified 2018-07

CONDITIONS: Infections, Streptococcal
Keywords: Booster vaccination; Pneumococcal vaccine; Catch-up vaccination; Pneumococcal disease; Safety; Immunogenicity
MeSH Terms: conditions — Streptococcal Infections; Pneumococcal Infections

ARMS (2):
- Pn-Pn group (Experimental): subjects from the Pn-Pn group, previously vaccinated with pneumococcal conjugate vaccine GSK1024850A in the Malian centre of study NCT00678301, receiving a booster dose of pneumococcal conjugate vaccine GSK1024850A
  Interventions: Biological: Pneumococcal vaccine GSK1024850A
- Zil-Pn group (Experimental): subjects from the unprimed group of the NCT00678301 Malian study centre, not previously vaccinated with any pneumococcal vaccine, receiving two doses of pneumococcal conjugate vaccine GSK1024850A
  Interventions: Biological: Pneumococcal vaccine GSK1024850A

INTERVENTIONS:
Biological: Pneumococcal vaccine GSK1024850A — Intramuscular injection, 1 or 2 doses

SUMMARY:
The purpose of this trial is to assess the safety, reactogenicity and immunogenicity of GSK Biologicals' pneumococcal conjugate vaccine GSK1024850A when administered either as a booster dose or as a two dose catch-up vaccination in the second year of life to the Malian subjects previously enrolled in the primary vaccination study NCT00678301.

This protocol posting deals with objectives & outcome measures of the booster phase. The objectives & outcome measures of the primary phase are presented in a separate protocol posting (NCT number = NCT00678301).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parent(s)/Legally Acceptable Representative(s) (LAR(s)) can and will comply with the requirements of the protocol.
* A male or female, between and including 15-21 months of age at the time of visit 1.
* For the Pn-Pn group, subjects who completed the full vaccination course in study NCT00678301. For the Zil-Pn group, subjects who were previously enrolled in the control group of study NCT00678301.
* Written informed consent, signed or thumb printed, obtained from the parent(s)/LAR(s) of the subject. Where parent(s)/LAR(s) are illiterate, the consent form will be countersigned by a witness.
* Healthy subjects as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s)/product(s) within 30 days preceding the first dose of vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to vaccination.
* Planned administration/administration of a vaccine not foreseen by the study protocol during the period starting from 30 days before each dose of study vaccine and ending 30 days after. Locally recommended vaccines for example Oral Polio Vaccine or influenza vaccine are always allowed, even if concomitantly administered with the study vaccines, but should be documented in the CRF.
* Concurrently participating in another clinical study at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Administration of any pneumococcal vaccine since the end of study NCT00678301.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, since the end of study NCT00678301, based on medical history and physical examination.
* Major congenital defects or serious chronic illness.
* History of any progressive neurological disorders or seizures.
* Acute disease and/or fever at the time of enrolment.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
* Administration of immunoglobulins and/or any blood products less than 3 months prior to visit 1 or planned use during the study.
* Child in care.

Ages: 15 Months to 21 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 218 (Actual)
Dates: Start 2009-11-12 (Actual); Primary Completion 2010-06-26 (Actual); Study Completion 2010-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Bamako, Mali

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Dicko A, Santara G, Mahamar A, Sidibe Y, Barry A, Dicko Y, Diallo A, Dolo A, Doumbo O, Shafi F, Francois N, Strezova A, Borys D, Schuerman L. Safety, reactogenicity and immunogenicity of a booster dose of the 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) in Malian children. Hum Vaccin Immunother. 2013 Feb;9(2):382-8. doi: 10.4161/hv.22692. Epub 2013 Jan 4. PMID 23291945
- [Background] Dicko A et al. Safety and immunogenicity of booster vaccination with 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) in Malian children. Abstract presented at the 7th World Congress of the World Society for Pediatric Infectious Diseases (WSPID). Melbourne, Australia, 16-19 November 2011 (Abstract 532).
- [Background] Dicko et al. Safety/reactogenicity and immunogenicity of 2-dose catch-up vaccination with 10-valent pneumococcal non-typeable Haemophilus influenzae protein-D conjugate vaccine (PHiD-CV) in Malian children. Abstract presented at the 8th International Symposium on Pneumococci & Pneumococcal Diseases (ISPPD), Iguaçu Falls, Brazil, 11-15 March 2012 (Abstract 085).
- [Derived] Dicko A, Dicko Y, Barry A, Sidibe Y, Mahamar A, Santara G, Dolo A, Diallo A, Doumbo O, Shafi F, Francois N, Yarzabal JP, Strezova A, Borys D, Schuerman L. Safety, reactogenicity and immunogenicity of 2-dose catch-up vaccination with 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) in Malian children in the second year of life: Results from an open study. Hum Vaccin Immunother. 2015;11(9):2207-14. doi: 10.1080/21645515.2015.1016679. PMID 26020101
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 113166 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 113166 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 113166 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 113166 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 113166 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 113166 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 113166 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 218 subjects were enrolled (147 subjects in the Synflorix Primed Group and 71 subjects in the Synflorix Unprimed Group). A total of 210 subjects were vaccinated in the booster vaccination study (141 out of 160 from the Synflorix Primed Group and 69 out of 78 from the Synflorix Unprimed Group).
Groups:
- Synflorix Primed Group: Subjects who were previously primed with the Synflorix™ vaccine in study 10PN-PD-DIT-032, received a booster dose of the Synflorix™ vaccine, administered intramuscularly in the thigh or deltoid, at 15-21 months of age (Study Month 0).
- Synflorix Unprimed Group: Unprimed subjects from the control group of study 10PN-PD-DIT-032, received a two dose catch-up vaccination with the Synflorix™ vaccine, administered intramuscularly in the thigh or deltoid, during the second year of life (at 15-21 months of age [Study Month 0] and at 17-23 months of age [Study Month 2]).
Period: Overall Study
Arm/Group | Synflorix Primed Group | Synflorix Unprimed Group
Started | 141 | 69
Completed | 140 | 66
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Considered to be part of the other group | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Synflorix Primed Group | Synflorix Unprimed Group | Total
Number analyzed (Participants) | 141 | 69 | 210
Age, Continuous [Mean (Standard Deviation); unit: Months] | 17 (1.11) | 16.9 (1.16) | 16.97 (1.12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 75 | 35 | 110
  Male | 66 | 34 | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Grade 3 Adverse Events (Solicited and Unsolicited)
Description: The incidence and nature of Grade 3 symptoms (solicited and unsolicited), reported during the 31-day (Days 0-30) post-vaccination are presented.
Time Frame: Within 31 days (Day 0-Day 30) after booster vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with at least one vaccine dose administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix Primed Group
Number analyzed (Participants) | 141
Participants
  Any symptom | 3
  General symptoms | 1
  Local symptoms | 2

2. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 30 millimeters (mm) of injection site.
Time Frame: Within 4 days (Day 0-Day 3) after the booster dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix Primed Group
Number analyzed (Participants) | 141
Participants
  Any Pain | 40
  Grade 3 Pain | 0
  Any Redness | 17
  Grade 3 Redness | 2
  Any Swelling | 67
  Grade 3 Swelling | 0

3. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were drowsiness, fatigue, fever [defined as axillary temperature equal to or above 37.5 degrees Celsius (°C)], irritability and loss of appetite. Any = occurrence of the symptom regardless of intensity grade. Grade 3 Drowsiness and Irritability = symptom that prevented normal activity. Grade 3 Loss of appetite = not eating at all. Grade 3 fever = fever > 39.5 °C. Related = symptom assessed by the investigator as related to the vaccination.
Time Frame: Within 4 days (Day 0-Day 3) after the booster dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix Primed Group
Number analyzed (Participants) | 141
Participants
  Any Drowsiness | 0
  Grade 3 Drowsiness | 0
  Related Drowsiness | 0
  Any Fever | 34
  Grade 3 Fever | 0
  Related Fever | 31
  Any Irritability | 8
  Grade 3 Irritability | 0
  Related Irritability | 8
  Any Loss of appetite | 1
  Grade 3 Loss of appetite | 0
  Related Loss of appetite | 1

4. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: as for outcome 2
Time Frame: Within 4 days (Day 0-Day 3) after each vaccine dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix Unprimed Group
Number analyzed (Participants) | 69
Participants
  Any Pain, Dose 1 | 22
  Grade 3 Pain, Dose 1 | 0
  Any Redness, Dose 1 | 6
  Grade 3 Redness, Dose 1 | 0
  Any Swelling, Dose 1 | 46
  Grade 3 Swelling, Dose 1 | 1
  Any Pain, Dose 2: number analyzed (Participants) | 67
  Any Pain, Dose 2 | 7
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 67
  Grade 3 Pain, Dose 2 | 0
  Any Redness, Dose 2: number analyzed (Participants) | 67
  Any Redness, Dose 2 | 2
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 67
  Grade 3 Redness, Dose 2 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 67
  Any Swelling, Dose 2 | 31
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 67
  Grade 3 Swelling, Dose 2 | 0
  Any Pain, Across Doses | 25
  Grade 3 Pain, Across Doses | 0
  Any Redness, Across Doses | 8
  Grade 3 Redness, Across Doses | 0
  Any Swelling, Across Doses | 55
  Grade 3 Swelling, Across Doses | 1

5. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: as for outcome 3
Time Frame: Within 4 days (Day 0-Day 3) after each vaccine dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix Unprimed Group
Number analyzed (Participants) | 69
Participants
  Any Drowsiness, Dose 1 | 1
  Grade 3 Drowsiness, Dose 1 | 0
  Related Drowsiness, Dose 1 | 1
  Any Fever, Dose 1 | 21
  Grade 3 Fever, Dose 1 | 0
  Related Fever, Dose 1 | 19
  Any Irritability, Dose 1 | 3
  Grade 3 Irritability, Dose 1 | 0
  Related Irritability, Dose 1 | 3
  Any Loss of appetite, Dose 1 | 1
  Grade 3 Loss of appetite, Dose 1 | 0
  Related Loss of appetite, Dose 1 | 0
  Any Drowsiness, Dose 2: number analyzed (Participants) | 67
  Any Drowsiness, Dose 2 | 0
  Grade 3 Drowsiness, Dose 2: number analyzed (Participants) | 67
  Grade 3 Drowsiness, Dose 2 | 0
  Related Drowsiness, Dose 2: number analyzed (Participants) | 67
  Related Drowsiness, Dose 2 | 0
  Any Fever, Dose 2: number analyzed (Participants) | 67
  Any Fever, Dose 2 | 17
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 67
  Grade 3 Fever, Dose 2 | 1
  Related Fever, Dose 2: number analyzed (Participants) | 67
  Related Fever, Dose 2 | 15
  Any Irritability, Dose 2: number analyzed (Participants) | 67
  Any Irritability, Dose 2 | 3
  Grade 3 Irritability, Dose 2: number analyzed (Participants) | 67
  Grade 3 Irritability, Dose 2 | 0
  Related Irritability, Dose 2: number analyzed (Participants) | 67
  Related Irritability, Dose 2 | 3
  Any Loss of appetite, Dose 2: number analyzed (Participants) | 67
  Any Loss of appetite, Dose 2 | 1
  Grade 3 Loss of appetite, Dose 2: number analyzed (Participants) | 67
  Grade 3 Loss of appetite, Dose 2 | 0
  Related Loss of appetite, Dose 2: number analyzed (Participants) | 67
  Related Loss of appetite, Dose 2 | 1
  Any Drowsiness, Across Doses | 1
  Grade 3 Drowsiness, Across Doses | 0
  Related Drowsiness, Across Doses | 1
  Any Fever, Across Doses | 34
  Grade 3 Fever, Across Doses | 1
  Related Fever, Across Doses | 30
  Any Irritability, Across Doses | 6
  Grade 3 Irritability, Across Doses | 0
  Related Irritability, Across Doses | 6
  Any Loss of appetite, Across Doses | 2
  Grade 3 Loss of appetite, Across Doses | 0
  Related Loss of appetite, Across Doses | 1

6. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: Within 31 days (Day 0-Day 30) after each vaccine dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix Primed Group | Synflorix Unprimed Group
Number analyzed (Participants) | 141 | 69
Participants | 95 | 57

7. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From the first vaccination up to one month (31 days) after the last vaccination for each subject
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Synflorix Primed Group | Synflorix Unprimed Group
Number analyzed (Participants) | 141 | 69
Participants | 0 | 0

8. Secondary Outcome: Concentrations of Antibodies Against Vaccine Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F
Description: Vaccine pneumococcal serotypes assessed were serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F. Concentrations were expressed as geometric mean concentrations (GMCs) in microgram per milliliter (μg/mL). Pneumococcal serotype specific total immunoglobuline G (IgG) antibodies were measured by 22F-inhibition Enzyme-linked immunosorbent assay (ELISA). The cut-off of the assay was ≥ 0.05 μg/mL.
Time Frame: Prior to (PRE) and one month after (POST) the booster immunization in the Synflorix Primed Group and prior to (PRE) the first dose and one month after (POST) the second dose of the catch-up vaccination in the Synflorix Unprimed Group
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects (i.e. those meeting all eligibility criteria, complying with the procedures and intervals defined in the protocol, with no elimination criteria during the study) for whom immunogenicity data were available.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix Primed Group | Synflorix Unprimed Group
Number analyzed (Participants) | 140 | 59
μg/mL
  Anti-1, PRE | 0.28 [0.23 to 0.35] | 0.04 [0.03 to 0.05]
  Anti-1, POST: number analyzed (Participants) | 139 | 57
  Anti-1, POST | 5.85 [5.07 to 6.76] | 3.2 [2.68 to 3.84]
  Anti-4, PRE | 0.32 [0.26 to 0.38] | 0.06 [0.04 to 0.09]
  Anti-4, POST: number analyzed (Participants) | 139 | 57
  Anti-4, POST | 10.44 [9.31 to 11.71] | 6.54 [5.47 to 7.82]
  Anti-5, PRE | 0.37 [0.32 to 0.43] | 0.04 [0.03 to 0.05]
  Anti-5, POST: number analyzed (Participants) | 139 | 57
  Anti-5, POST | 6.07 [5.2 to 7.1] | 3.05 [2.4 to 3.87]
  Anti-6B, PRE | 0.66 [0.55 to 0.8] | 0.03 [0.03 to 0.04]
  Anti-6B, POST: number analyzed (Participants) | 139 | 57
  Anti-6B, POST | 4.44 [3.69 to 5.33] | 0.78 [0.57 to 1.08]
  Anti-7F, PRE | 0.68 [0.59 to 0.8] | 0.04 [0.03 to 0.06]
  Anti-7F, POST: number analyzed (Participants) | 139 | 57
  Anti-7F, POST | 7.82 [6.92 to 8.85] | 4.5 [3.8 to 5.33]
  Anti-9V, PRE | 0.73 [0.61 to 0.87] | 0.03 [0.03 to 0.04]
  Anti-9V, POST: number analyzed (Participants) | 139 | 57
  Anti-9V, POST | 7.99 [6.86 to 9.3] | 1.48 [1.2 to 1.83]
  Anti-14, PRE | 0.9 [0.73 to 1.09] | 0.11 [0.09 to 0.14]
  Anti-14, POST: number analyzed (Participants) | 139 | 57
  Anti-14, POST | 9.75 [8.02 to 11.85] | 4.51 [3.63 to 5.61]
  Anti-18C, PRE | 0.92 [0.79 to 1.07] | 0.05 [0.04 to 0.07]
  Anti-18C, POST: number analyzed (Participants) | 139 | 57
  Anti-18C, POST | 23.99 [20.29 to 28.37] | 10.95 [8.5 to 14.1]
  Anti-19F, PRE | 0.82 [0.66 to 1.04] | 0.09 [0.06 to 0.14]
  Anti-19F, POST: number analyzed (Participants) | 139 | 57
  Anti-19F, POST | 12.96 [10.96 to 15.34] | 8.52 [5.58 to 13]
  Anti-23F, PRE | 0.35 [0.28 to 0.45] | 0.03 [0.03 to 0.04]
  Anti-23F, POST: number analyzed (Participants) | 139 | 57
  Anti-23F, POST | 4.25 [3.54 to 5.11] | 1.05 [0.74 to 1.49]

9. Secondary Outcome: Opsonophagocytic Activity Against Pneumococcal Serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F
Description: OPA titers against pneumococcal serotypes 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F and 23F (Opsono-1, -4, -5, -6B, -7F, -9V, -14, -18C, -19F and -23F) were calculated, expressed as geometric mean titers (GMTs) and tabulated. The seropositivity cut-off for the assay was ≥ 8.
Time Frame: as for outcome 8
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects (i.e. those meeting all eligibility criteria, complying with the procedures and intervals defined in the protocol, with no elimination criteria during the study) for whom immunogenicity data were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix Primed Group | Synflorix Unprimed Group
Number analyzed (Participants) | 139 | 58
Titers
  Opsono-1, PRE | 9.3 [7.3 to 11.8] | 5.8 [4.3 to 7.8]
  Opsono-1, POST: number analyzed (Participants) | 139 | 57
  Opsono-1, POST | 661.7 [513.5 to 852.6] | 108.7 [79.5 to 148.6]
  Opsono-4, PRE: number analyzed (Participants) | 139 | 57
  Opsono-4, PRE | 24 [16.7 to 34.6] | 11.8 [6.3 to 22.1]
  Opsono-4, POST: number analyzed (Participants) | 139 | 55
  Opsono-4, POST | 6541.7 [5468.5 to 7825.6] | 2716.7 [2149 to 3434.2]
  Opsono-5, PRE: number analyzed (Participants) | 133 | 58
  Opsono-5, PRE | 9 [7.4 to 10.9] | 4.3 [3.7 to 5]
  Opsono-5, POST: number analyzed (Participants) | 139 | 57
  Opsono-5, POST | 340.5 [272.2 to 426] | 71.9 [51.8 to 99.7]
  Opsono-6B, PRE: number analyzed (Participants) | 116 | 46
  Opsono-6B, PRE | 82.6 [50.5 to 135.1] | 38.7 [16.2 to 92]
  Opsono-6B, POST: number analyzed (Participants) | 134 | 50
  Opsono-6B, POST | 1729 [1361.9 to 2194.9] | 1202.9 [701.3 to 2063]
  Opsono-7F, PRE: number analyzed (Participants) | 133 | 51
  Opsono-7F, PRE | 3230.6 [2588.4 to 4032.1] | 2454.4 [1587.3 to 3795.1]
  Opsono-7F, POST: number analyzed (Participants) | 136 | 57
  Opsono-7F, POST | 9116.9 [7679.8 to 10822.9] | 9161.1 [7254.1 to 11569.4]
  Opsono-9V, PRE: number analyzed (Participants) | 100 | 44
  Opsono-9V, PRE | 407.9 [265.3 to 627] | 138.2 [63.2 to 302.6]
  Opsono-9V, POST: number analyzed (Participants) | 111 | 43
  Opsono-9V, POST | 3640.4 [2859 to 4635.3] | 4596.5 [3519.4 to 6003.3]
  Opsono-14, PRE: number analyzed (Participants) | 112 | 36
  Opsono-14, PRE | 84.3 [53.4 to 132.9] | 18.8 [8.4 to 42.3]
  Opsono-14, POST: number analyzed (Participants) | 109 | 41
  Opsono-14, POST | 3281.8 [2488.4 to 4328.2] | 2246.1 [1621.5 to 3111.1]
  Opsono-18C, PRE: number analyzed (Participants) | 95 | 33
  Opsono-18C, PRE | 6 [4.8 to 7.5] | 6.4 [4 to 10.3]
  Opsono-18C, POST: number analyzed (Participants) | 106 | 38
  Opsono-18C, POST | 2413.2 [1925.5 to 3024.6] | 2045.3 [1161.5 to 3601.8]
  Opsono-19F, PRE: number analyzed (Participants) | 124 | 57
  Opsono-19F, PRE | 12.8 [9.3 to 17.7] | 4.8 [3.7 to 6.3]
  Opsono-19F, POST: number analyzed (Participants) | 127 | 47
  Opsono-19F, POST | 1084.2 [828.9 to 1418.1] | 693.7 [350.8 to 1371.6]
  Opsono-23F, PRE: number analyzed (Participants) | 132 | 49
  Opsono-23F, PRE | 90.7 [52.7 to 156.2] | 30.4 [12.9 to 71.4]
  Opsono-23F, POST: number analyzed (Participants) | 137 | 57
  Opsono-23F, POST | 3476.4 [2706.8 to 4464.7] | 3571 [2793.4 to 4565.1]

10. Secondary Outcome: Concentrations of Antibodies Against Cross-reactive Pneumococcal Serotypes 6A and 19A
Description: Cross-reactive pneumococcal serotypes assessed were serotypes 6A and 19A. Concentrations were expressed as geometric mean concentrations (GMCs) in microgram per milliliter (μg/mL). The antibody concentrations against the cross-reactive pneumococcal serotypes 6A and 19A were determined by 22F-inhibition Enzyme-linked immunosorbent assay (ELISA). The cut-off of the assay was ≥ 0.05 μg/mL.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Synflorix Primed Group | Synflorix Unprimed Group
Number analyzed (Participants) | 140 | 59
μg/mL
  Anti-6A, PRE | 0.13 [0.11 to 0.17] | 0.04 [0.03 to 0.05]
  Anti-6A, POST: number analyzed (Participants) | 139 | 57
  Anti-6A, POST | 0.55 [0.42 to 0.73] | 0.1 [0.07 to 0.14]
  Anti-19A, PRE: number analyzed (Participants) | 140 | 58
  Anti-19A, PRE | 0.16 [0.13 to 0.22] | 0.06 [0.04 to 0.09]
  Anti-19A, POST: number analyzed (Participants) | 130 | 57
  Anti-19A, POST | 1.13 [0.83 to 1.53] | 1.36 [0.91 to 2.03]

11. Secondary Outcome: Opsonophagocytic Activity Against Cross-reactive Pneumococcal Serotypes 6A and 19A
Description: OPA titers against pneumococcal serotypes 6A and 19A (Opsono-6A and Opsono-19A) were calculated, expressed as geometric mean titers (GMTs) and tabulated. The seropositivity cut-off for the assay was ≥ 8.
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Synflorix Primed Group | Synflorix Unprimed Group
Number analyzed (Participants) | 138 | 58
Titers
  Opsono-6A, PRE: number analyzed (Participants) | 127 | 54
  Opsono-6A, PRE | 18.7 [12.2 to 28.6] | 24 [12.5 to 46.3]
  Opsono-6A, POST: number analyzed (Participants) | 126 | 48
  Opsono-6A, POST | 100.7 [60.4 to 168] | 106.3 [46.3 to 244]
  Opsono-19A, PRE | 6.2 [5.1 to 7.6] | 5.9 [4.2 to 8.3]
  Opsono-19A, POST: number analyzed (Participants) | 134 | 54
  Opsono-19A, POST | 91.5 [60.4 to 138.5] | 171.2 [94.2 to 311.3]

12. Secondary Outcome: Concentrations of Antibodies Against Protein D (PD)
Description: Concentrations of antibodies against protein D (PD) were determined by ELISA assay. Concentrations were expressed as geometric mean concentrations (GMCs) in ELISA units per milliliter (EL.U/mL). Concentration of specific PD antibodies was determined, using a standard reference serum. The cut-off of the assay is ≥ 100 ELISA units per milliliter (EL.U/mL).
Time Frame: as for outcome 8
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Synflorix Primed Group | Synflorix Unprimed Group
Number analyzed (Participants) | 139 | 59
EL.U/mL
  Anti-PD, PRE | 301.1 [257.7 to 351.8] | 62.1 [54.9 to 70.3]
  Anti-PD, POST: number analyzed (Participants) | 139 | 56
  Anti-PD, POST | 3710.1 [3109 to 4427.4] | 839.3 [643.5 to 1094.6]

ADVERSE EVENTS:
Time Frame: Solicited AEs: within 4 days (Day 0-Day 3) after each vaccine dose; Unsolicited AEs: within 31 days (Day 0-Day 30) after each vaccine dose; SAEs: from the first vaccination up to one month (31 days) after the last vaccination for each subject.
Arm/Group | Synflorix Primed Group | Synflorix Unprimed Group
Serious Adverse Events (participants affected / at risk) | 0/141 | 0/69
Other Adverse Events (participants affected / at risk) | 125/141 | 64/69
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Synflorix Primed Group (N=141) | Synflorix Unprimed Group (N=69)
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 38 (41) | 22 (25)
Circumcision (Surgical and medical procedures) | 1 (1) | 4 (4)
Enteritis (Gastrointestinal disorders) | 6 (6) | 8 (10)
Erythema (Skin and subcutaneous tissue disorders) | 17 (17) | 8 (8)
Gastroenteritis (Infections and infestations) | 12 (12) | 15 (16)
Injection site induration (General disorders) | 5 (5) | 10 (10)
Irritability (Psychiatric disorders) | 8 (8) | 6 (6)
Pain (General disorders) | 40 (40) | 25 (29)
Pyrexia (General disorders) | 34 (35) | 34 (38)
Rhinitis (Infections and infestations) | 26 (27) | 14 (15)
Skin infection (Infections and infestations) | 9 (9) | 3 (3)
Swelling (General disorders) | 67 (67) | 55 (77)
Wound (Injury, poisoning and procedural complications) | 1 (1) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.